CLINICAL TRIAL: NCT03052062
Title: Lipidrive Dietary Supplement Tolerance Study Based on Blood, Urine, and Hemodynamic Biological Parameters.
Brief Title: Tolerance Study of the Dietary Supplement Lipidrive (ECPH1-03)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Valbiotis (Industry)
Collaborators: University Hospital, Clermont-Ferrand (Other); Université Blaise Pascal, Clermont-Ferrand (Other); Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01187-44
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lipidrive (Experimental): Dose 1 : 2,6 g (4 capsules) Lipidrive per day during 12 weeks Dose 2 : 5,2 g (8 capsules) Lipidrive per day during 12 weeks, 2 weeks (wash-out period) between the 2 doses
  Interventions: Dietary Supplement: Lipidrive

INTERVENTIONS:
Dietary Supplement: Lipidrive — LipiDrive, 4 to 8 capsules per day, oral administration. Dose 1: 2.6 g Lipidrive per day Dose 2: 5.2 g Lipidrive per day

SUMMARY:
The objectives of this clinical study are to determine the tolerance of dietary supplement Lipidrive through the evaluation of several parameters :

* Various blood biological parameters
* Urinary parameters
* Hemodynamic indicators
* Cardiac function
* Anthropometric variables

DETAILED DESCRIPTION:
Primary objectives of this study :

Evaluate the effects of two doses of the product on:

* Various blood biological parameters for tolerance (preprandial): blood glucose, insulin, HOMA-IR, glycated hemoglobin, fructosamine, total cholesterol, triglycerides, HDL-cholesterol, LDL-cholesterol, oxidized LDL, us-CRP, creatinine, ASAT, ALAT, gGT, alkaline phosphatase, bilirubin, urea.
* Urinary parameters: urea, creatinine.
* Hemodynamic indicators: heart rate and blood pressure.
* Cardiac function: ECG.
* Anthropometric variables: weight, waist, hips, waist/hip ratio, body composition using bioelectric impendence analysis.

Secondary objectives of this study:

Evaluate the effects of the highest dose on:

- Adiponectin, leptin, TNF-α, and the evolution kinetics of blood glucose and blood insulin levels following a standard breakfast, with or without the acute administration of the Lipidrive dietary supplement.

Two questionnaires (one on eating habits over 3 days and another on physical and sports activities) will be completed at various times (cf. below). A "satisfaction" questionnaire will also be completed at the end of the study.

A serum bank will be created (ghrelin, resistin, GIP, GLP-1, IL-6, IL-1 beta, CCK), and stools will be collected at V2 and V5 for subsequent microbiota analysis (aliquoting performed by the AME2P laboratory, which will send the samples to BIOFORTIS Nantes at the end of the trial).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 45 to 65 years (inclusive)
* BMI between 30 kg/m² (inclusive) and 40 kg/m² (non-inclusive) and/or a waist/hips ratio > 0.9
* Non-smoker or smokes maximum 10 cigarettes per day
* Stable weight for at least 3 months before the start of the study
* Regular physical activity for 3 months before the start of the study, subject agreeing to maintain this level of activity over the course of the study
* Stable eating habits for 3 months before the start of the study, subject agreeing to maintain these eating habits over the course of the study
* Willing and able to comply with the protocol, subject agreeing to give their informed written consent
* Registered with a social security scheme
* Subject agreeing to be registered in the national directory of volunteers participating in biomedical research

Following the biological screening conducted during the inclusion visit, run-in subjects will be included at the following visit according to the following criteria:

* FBC with no clinically significant anomalies according to the investigator
* ASAT ≤ 1.55 μkat/L or ≤ 92 U/L
* ALAT ≤ 1.7 μkat/L or ≤ 101 U/L
* gGT ≤ 2.55 μkat/L or ≤ 152 U/L
* 45 ≤ Creatinine ≤ 104 μmol/L (± 10%)
* Total bilirubin < 17.1 μmol/L (± 10%)
* 1.7 mmol/L ≤ Urea ≤ 8.3 mmol/L (± 10%)
* us-CRP ≤ 5 mg/L (± 10%).

Exclusion Criteria:

* Confirmed or suspected food allergy to the test product (describe)
* Subject with chronic condition or specific circumstances that the investigator considers incompatible with participation in the study
* Subject taking anti-diabetic treatment
* Subject taking lipo-regulating (fibrates, statins, nicotinic acid) or anti-dyslipidemia drugs
* Subject consuming dietary supplements (V0 could be conducted at least 1 month after completely stopping the supplements)
* Subject consuming grapefruit or orange juice (enzyme inhibitor)
* Subject consuming food products supplemented with phytosterols, beta glucans, konjac, and/or cinnamon (V0 could be conducted at least 3 months after completely stopping the supplements) (list to be drawn up at the time of the study)
* Unstable blood pressure equal to or over 160/95
* Subject undergoing treatment that, according to the investigator, could interfere with the evaluation of the study criteria
* Subject who has been on a low-calorie diet in the 3 months prior to the study and/or intends to go on a diet during the study
* Subject with serious history of anorexia nervosa, bulimia or other eating disorders
* Vegetarian or vegan
* Extreme eating habits
* Subject participating in another clinical study or in an exclusion period following a previous clinical study
* Subject who has received over 4500 euros in compensation since the start of the calendar year (sum can vary according to regulations)
* Subject with a linguistic or physical incapacity to provide written informed consent
* Refusal to provide written consent
* Subject deprived of liberty by administrative or judicial order, under trusteeship or guardianship
* Subject who cannot be contacted by telephone in case of emergency

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Changes in fasting blood glucose | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in mmol/L
Changes in fasting blood glucose | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in mmol/L
Changes in fasting insulinemia | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline)) in mUI/L
Changes in fasting insulinemia | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in mUI/L
Changes in fasting HOMA-IR | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline)
Changes in fasting HOMA-IR | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks)
Changes in glycated hemoglobin | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in %
Changes in glycated hemoglobin | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in %
Changes in fasting fructosamin | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in µmol/L
Changes in fasting fructosamin | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in µmol/L
Changes in fasting total cholesterol | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in mmol/L
Changes in fasting total cholesterol | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in mmol/L
Changes in fasting HDL cholesterol | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in mmol/L
Changes in fasting HDL cholesterol | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in mmol/L
Changes in fasting LDL cholesterol | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in mmol/L
Changes in fasting LDL cholesterol | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in mmol/L
Changes in fasting triglycerides | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in mmol/L
Changes in fasting triglycerides | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in mmol/L
Changes in oxidized LDL | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in mmol/L
Changes in oxidized LDL | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in mmol/L
Changes in us-CRP | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in mg/L
Changes in us-CRP | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in mmol/L
Changes in blood creatinine | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in mg/dL
Changes in blood creatinine | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in mg/dL
Changes in fasting blood levels of ASAT (Aspartate aminotransferase) and ALAT (Alanine aminotransferase) | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in UI/L
Changes in fasting blood levels of ASAT (Aspartate aminotransferase) and ALAT (Alanine aminotransferase) | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in UI/L
Changes in fasting blood levels of GGT (Gamma glutamyltransferase) | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in UI/L
Changes in fasting blood levels of GGT (Gamma glutamyltransferase) | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in UI/L
Changes in fasting alkaline phosphatase | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in UI/L
Changes in fasting alkaline phosphatase | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in UI/L
Changes in fasting blood bilirubin | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in µmol/L
Changes in fasting blood bilirubin | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in µmol/L
Changes in fasting blood urea | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in mg/dL
Changes in fasting blood urea | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in mg/dL
Changes in heart rate | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in bpm
Changes in heart rate | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in bpm
Changes in SBP (systolic blood pressure) and DBP (diastolic blood pressure) | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in mmHg (mean of the two measures for each parameter at each visit)
Changes in SBP (systolic blood pressure) and DBP (diastolic blood pressure) | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in mmHg (mean of the two measures for each parameter at each visit)
Changes in cardiac function (electrocardiogram, ECG) | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline)
Changes in cardiac function (electrocardiogram, ECG) | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks)
Changes in body weight | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline) in kg
Changes in body weight | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks) in kg
Changes in WC (waist circumference) | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline)
Changes in WC (waist circumference) | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks)
Changes in HC (hip circumference) | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline)
Changes in HC (hip circumference) | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks)
Changes in WHR (waist to hip ratio) | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline)
Changes in WHR (waist to hip ratio) | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks)
Changes in body composition | 12 weeks
  Defined as the difference V3 (12 weeks) - V2 (baseline), using bioelectric impendence analysis
Changes in body composition | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks), using bioelectric impendence analysis

SECONDARY OUTCOMES:
Changes in fasting blood adiponectin | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks)
Changes in fasting blood leptin | 26 weeks
  Defined as the difference V5 (26 weeks) - V4 (14 weeks)
Changes in the evolution of glycemia during an oral glucid tolerance test | 26 weeks
  Changes between V5 (26 weeks) and V4 (14 weeks) visits (defined as the difference V4-V3 in mmol/L) of glycemia at 15, 30, 45, 60, 90 and 120 minutes between T0 and T120 minutes following a standard breakfast and considering the following time-points: T-10, T-5, T0, T15, T30, T45, T60, T90 and T120
Changes in the incremental area under the curve (glycemia response) during an oral glucid tolerance test | 26 weeks
  Changes between V5 (26 weeks) and V4 (14 weeks) visits (defined as the difference V4-V3 in mmol/L) of incremental Area Under the Curve (iAUC) of glycemia between T0 and T120 minutes following a standard breakfast (iAUC0-120min) and considering the following time-points: T-10, T-5, T0, T15, T30, T45, T60, T90 and T120
Changes in the glycemia Cmax during an oral glucid tolerance test | 26 weeks
  Changes between V5 (26 weeks) and V4 (14 weeks) visits (defined as the difference V4-V3 in mUIl/L) of glycemia Cmax between T0 and T120 minutes following a standard breakfast and considering the following time-points: T-10, T-5, T0, T15, T30, T45, T60, T90 and T120
Changes in the glycemia Δpeak during an oral glucid tolerance test | 26 weeks
  Changes between V5 (26 weeks) and V4 (14 weeks) visits (defined as the difference V4-V3 in mmol/L) of Δpeak (difference from the baseline at Cmax), between T0 and T120 minutes following a standard breakfast and considering the following time-points: T-10, T-5, T0, T15, T30, T45, T60, T90 and T120
Changes in the evolution of insulinemia during an oral glucid tolerance test | 26 weeks
  Changes between V5 (26 weeks) and V4 (14 weeks) visits (defined as the difference V4-V3 in mUI/L) of insulinemia at 15, 30, 45, 60, 90 and 120 minutes between T0 and T120 minutes following a standard breakfast and considering the following time-points: T-10, T-5, T0, T15, T30, T45, T60, T90 and T120
Changes in the incremental area under the curve (insulinemia response) during an oral glucid tolerance test | 26 weeks
  Changes between V5 (26 weeks) and V4 (14 weeks) visits (defined as the difference V4-V3 in mUI/L) of incremental Area Under the Curve (iAUC) of insulinemia between T0 and T120 minutes following a standard breakfast (iAUC0-120min) and considering the following time-points: T-10, T-5, T0, T15, T30, T45, T60, T90 and T120
Changes in the insulinemia Cmax during an oral glucid tolerance test | 26 weeks
  Changes between V5 (26 weeks) and V4 (14 weeks) visits (defined as the difference V4-V3 in mUIl/L) of insulinemia Cmax between T0 and T120 minutes following a standard breakfast and considering the following time-points: T-10, T-5, T0, T15, T30, T45, T60, T90 and T120
Changes in the insulinemia Δpeak during an oral glucid tolerance test | 26 weeks
  Changes between V5 (26 weeks) and V4 (14 weeks) visits (defined as the difference V4-V3 in mUIl/L) of Δpeak (difference from the baseline at Cmax), between T0 and T120 minutes following a standard breakfast and considering the following time-points: T-10, T-5, T0, T15, T30, T45, T60, T90 and T120

OTHER OUTCOMES:
Changes in stools microbiota | 26 weeks
  Changes between V5 (26 weeks) and V4 (14 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, MD, PhD, Principal Investigator — Centre d'Investigation Clinique INSERM 501, Clermont-Ferrand, France; Sébastien Peltier, PhD, Study Director — Valbiotis
Locations (1):
- Centre d'Investigation Clinique, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Yes